CLINICAL TRIAL: NCT07331779
Title: Timing Matters: Comparing Pre , Peri , and Post Rehabilitation tDCS in Acute Stroke Recovery
Brief Title: Effect of tDCS Timing on Motor Recovery in Acute Stroke Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Bornheim Stephen, Prof., University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 45.482.838
Record Dates: First submitted 2025-12-26; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Active tDCS Before Rehabilitation (Experimental): Active tDCS Before Rehabilitation
  Interventions: Device: tDCS; Device: Sham Transcranial Direct Current Stimulation (Sham tDCS)
- Arm 2 - Active tDCS During Rehabilitation (Experimental): Active tDCS During Rehabilitation
  Interventions: Device: tDCS; Device: Sham Transcranial Direct Current Stimulation (Sham tDCS)
- Arm 3 - Active tDCS After Rehabilitation (Experimental): Active tDCS After Rehabilitation
  Interventions: Device: tDCS; Device: Sham Transcranial Direct Current Stimulation (Sham tDCS)

INTERVENTIONS:
Device: tDCS — Transcranial Direct Current Stimulation (tDCS) is delivered using a non-invasive electrical stimulation device that applies a low-intensity direct current (2 mA) through two saline-soaked sponge electrodes placed on the scalp. Each participant receives three stimulation sessions per day: one before, one during, and one after their rehabilitation session. In each randomized group, only one of these three daily stimulations is active, while the other two are sham (brief ramp-up and ramp-down without sustained current). The active stimulation lasts 20 minutes. Sham sessions mimic the initial sensations of stimulation to maintain blinding. Electrode placement is standardized according to the lesioned hemisphere. All participants receive five consecutive days of this combined protocol alongside their usual rehabilitation program.
  Other Names: Rehabilitation
Device: Sham Transcranial Direct Current Stimulation (Sham tDCS) — Sham tDCS is delivered using the same device and electrode placement as active stimulation, but without administering a sustained electrical current. The device applies a brief ramp-up and ramp-down of current at the beginning and end of the session to mimic the initial sensations of active tDCS (e.g., tingling or warmth), after which no current is delivered. Each participant receives three tDCS sessions per day (before, during, and after rehabilitation), but only one is active; the other two are sham. Sham stimulation is used to maintain double-blinding and ensure that participants and assessors cannot distinguish between active and inactive sessions.

SUMMARY:
This randomized, double-blind, sham-controlled clinical trial investigates how the timing of transcranial direct current stimulation (tDCS) influences functional recovery during acute stroke rehabilitation. Sixty hospitalized patients with confirmed acute stroke will be randomly assigned to one of three groups. Each day, all participants will receive three tDCS sessions: one before, one during, and one after their rehabilitation session. In each group, only one of these three daily stimulations is active, while the other two are sham, allowing a direct comparison of timing effects while maintaining blinding. All participants will complete five consecutive days of conventional rehabilitation combined with the tDCS protocol. Functional, sensory, psychological, and motor outcomes will be assessed at baseline and at the end of the intervention week. The study aims to determine whether the timing of tDCS application influences early post-stroke recovery and to inform the design of future confirmatory trials.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for stroke rehabilitation Hospitalized in a stroke rehabilitation unit at CHU de Liège.

Confirmed acute stroke Diagnosis of acute stroke (ischemic or hemorrhagic) confirmed by neuroimaging, according to local clinical practice.

Time since stroke In the acute/subacute phase, as defined in the protocol (e.g., within X days/weeks after stroke onset) - to be specified exactly as in your protocol.

Age Age ≥ 18 years.

Capacity to consent Able to understand the study information and provide written informed consent.

Motor impairment of the upper limb Presence of motor deficit of the upper limb on the affected side, sufficient to perform the WMFT tasks (according to protocol thresholds, if specified).

Medically stable Clinically stable and judged by the treating physician as able to participate in daily rehabilitation and tDCS sessions.

Exclusion Criteria:

* Contraindications to tDCS or cranial stimulation

Implanted electronic devices in the head or neck (e.g., deep brain stimulator, cochlear implant, implanted neurostimulator, pacemaker with leads near the head).

Metal implants in the skull (excluding dental fillings) in the area of stimulation.

Large skull defect or craniectomy over the stimulation site.

History of seizures History of epilepsy or unprovoked seizures not adequately controlled, if considered a contraindication to tDCS by the investigator.

Severe cognitive or communication impairment Severe cognitive impairment, aphasia, or comprehension difficulties preventing understanding of the study or execution of the tasks, as judged by the investigator.

Severe comorbidities Unstable medical conditions (e.g., uncontrolled cardiac, respiratory, metabolic, or systemic disease) that could interfere with participation or increase risk.

Severe psychiatric disorder Current severe psychiatric illness (e.g., psychosis, severe untreated major depression) that may affect cooperation or safety, as judged by the investigator.

Skin conditions at electrode sites Skin lesions, infections, severe dermatitis, or wounds at or near the planned electrode placement sites.

Concurrent participation in another interventional trial Participation in another interventional clinical trial that could interfere with the outcomes or safety of this study.

Pregnancy Pregnancy or breastfeeding, if considered a contraindication according to local tDCS safety policy (optional, depending on your protocol stance).

Any other reason Any condition or circumstance that, in the opinion of the investigator, makes the patient unsuitable for the study or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in upper limb motor function (Wolf Motor Function Test, WMFT) | Baseline (Day 1, pre-intervention) to end of intervention (Day 5, post-intervention).
  The WMFT assesses upper limb motor function using timed and functional tasks. The primary outcome is the change in WMFT performance (time and/or functional score) between baseline and Day 5, comparing the three timing conditions of active tDCS (before, during, after rehabilitation).
  The Wolf Motor Function Test (WMFT) will be used to assess upper-limb motor performance. The Functional Ability Scale ranges from 0 to 5, with higher scores indicating better functional movement quality. Performance Time is measured from 0 to 120 seconds, with lower times indicating better performance.

SECONDARY OUTCOMES:
Change in sensory function (Semmes-Weinstein Monofilament Test, SWMT) | Baseline (Day 1) to Day 5.
  The SWMT evaluates cutaneous sensory thresholds using calibrated monofilaments. The outcome is the change in sensory detection thresholds between baseline and Day 5.
  The Semmes-Weinstein Monofilament Test will be used to assess cutaneous pressure sensitivity. Monofilaments range from approximately 0.008 g to 300 g. Lower detectable force values indicate better tactile sensitivity, whereas higher detectable force values indicate worse sensory function.
Change in spasticity (Tardieu Scale) | Baseline (Day 1) to Day 5.
  The Tardieu Scale assesses spasticity by measuring muscle reaction to passive stretch at different velocities. The outcome is the change in Tardieu scores (e.g., angle of catch, quality of muscle reaction) between baseline and Day 5.
  The Tardieu Spasticity Scale will be used to assess spasticity. It includes two components: (1) the Quality of Muscle Reaction score (0-4, where higher scores indicate worse spasticity), and (2) the Angle of Muscle Reaction, measured in degrees from 0° to the joint's full passive range, where higher values indicate a better outcome.
Change in functional independence (Barthel Index) | Baseline (Day 1) to Day 5.
  The Barthel Index measures independence in activities of daily living. The outcome is the change in total Barthel score between baseline and Day 5.
  "The Barthel Index of Activities of Daily Living will be used to assess functional independence. Scores range from 0 to 100, with higher scores indicating better independence and lower scores indicating greater dependency.
Change in balance and gait (Tinetti Performance-Oriented Mobility Assessment) | Baseline (Day 1) to Day 5.
  The Tinetti test evaluates balance and gait performance and estimates fall risk. The outcome is the change in Tinetti total score between baseline and Day 5.
  The Tinetti Assessment Tool (Performance-Oriented Mobility Assessment) will be used to evaluate balance and gait. The Balance Subscale ranges from 0 to 16 and the Gait Subscale from 0 to 12. The total score ranges from 0 to 28. In all cases, higher scores indicate better performance and lower fall risk.
Change in health-related quality of life after stroke (Stroke Impact Scale, SIS) | Baseline (Day 1) to Day 5.
  The Stroke Impact Scale is a patient-reported questionnaire assessing multiple domains affected by stroke (e.g., physical function, emotion, participation). The outcome is the change in SIS scores between baseline and Day 5.
  The Stroke Impact Scale (Version 3.0) will be used to assess patient-reported impact of stroke across multiple functional domains. Items are scored from 1 to 5, with higher scores indicating better perceived function. Domain scores are transformed to a 0-100 scale, where higher values indicate better outcomes.
Change in anxiety and depression (Hospital Anxiety and Depression Scale, HADS) | Baseline (Day 1) to Day 5.
  The HADS evaluates symptoms of anxiety and depression using a 14-item questionnaire. The outcome is the change in anxiety and depression subscale scores between baseline and Day 5.
  "The Hospital Anxiety and Depression Scale will be used to assess symptoms of anxiety and depression. Each subscale ranges from 0 to 21, with higher scores indicating worse symptoms. The optional total score ranges from 0 to 42, with higher values indicating greater emotional distress.
Incidence of adverse events and tolerability of tDCS | Throughout the 5 days of intervention.
  Number, type, and severity of adverse events potentially related to tDCS (e.g., headache, skin irritation, discomfort, dizziness) recorded at each session using standardized questioning and observation.

IPD SHARING:
Plan to Share IPD: No